CLINICAL TRIAL: NCT03459508
Title: Ocular Findings in Women With Primary Antiphospholipid Syndrome and Their Association to Bad Obstetric Outcome
Brief Title: Ocular Findings in Women With Primary Antiphospholipid Syndrome
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed AA Wali, MD, Lecturer of Obstetrics and Gynecology, Cairo University
Other Study IDs: N-2aa5-2018
Record Dates: First submitted 2018-02-22; First posted 2018-03-09 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Primary Antiphospholipid Syndrome
Keywords: Antiphospholipid Syndrome - Bad obstetric history - Ocular
MeSH Terms: interventions — Slit Lamp Microscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Primary antiphospholipid syndrome women: 1. Informed consent
  2. Detailed history emphasizing on
     a. obstetric complications related to antiphospholipid syndrome: i. Recurrent miscarriage ii. Fetal demise iii. Fetal growth restriction iv. Severe pre-eclampsia or eclampsia v. Placental insufficiency vi. Placental abruption b. Systemic vascular complications related to antiphospholipid syndrome: i. Arterial thrombosis ii. Venous thrombosis iii. Small-vessel thrombosis
  3. Revision of diagnosis of primary antiphospholipid syndrome:
  4. Exclusion of antiphospholipid syndrome secondary to SLE and other autoimmune diseases by: antinuclear (ANA), anti-Smith (Sm) and anti-double stranded DNA (dsDNA) antibodies.
  5. Ophthalmological examination:
  Interventions: Diagnostic Test: Ophthalmological examination

INTERVENTIONS:
Diagnostic Test: Ophthalmological examination — Detailed anterior segment examination using slit-lamp biomicroscopy for signs of anterior uveitis, and detailed fundus examination using slit-lamp fundus biomicroscopy with + 90 diopter lens searching for signs of vasculitis and posterior uveitis.
  Other Names: slit lamp biomicroscopy; slit lamp exam

SUMMARY:
Antiphospholipid antibody syndrome (APS) is an autoimmune disease characterized by systemic thrombosis and bad obstetric history. APS secondary to another medical disorder is the most common. Visual and ocular changes e.g. vaso-occlusive disease of retinal and choroidal vessels are found in patients with secondary APS. Patients with primary APS have also been reported to have ocular changes e.g. retinal vascular occlusion

The aim of our study to detect prevalence of ocular changes in women diagnosed with primary APS and correlation of these changes with adverse obstetric outcome. If a correlation is present, ocular findings in women with APS could be used in the future as a predictor for poor obstetric outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 35 years
* Females with primary antiphospholipid syndrome

Exclusion Criteria:

* Age: below 18 years and above 35 years
* Auto-immune diseases e.g. SLE and other connective tissue disease
* Medical diseases causing retinal vascular changes e.g. hypertension, diabetes mellitus, sickle cell anemia.
* Previous vitreo-retinal surgery

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients (inpatient or outpatient) with primary antiphospholipid syndrome at Kasr-Alainy hospital (The Cairo University Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
The incidence of Ocular changes in females with antiphospholipid syndrome | On the same day of enrollment into the study
  Number of participants with ocular findings detected by ophthalmological examination

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AA Wali, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided